CLINICAL TRIAL: NCT02606110
Title: Pilot Study Investigating the Use of the ReBuilder to Treat Chemotherapy Induced Peripheral Neuropathy in Patients With Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: PI decided no longer to pursue
Sponsor: Eastern Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ERMC 14-11
Record Dates: First submitted 2015-05-26; First posted 2015-11-17 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Peripheral Neuropathy
Keywords: ReBuilder; breast cancer; chemotherapy induced
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate the effect of the ReBuilder in the treatment of individuals with breast cancer and chemotherapy induced peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer referred to Physical Therapy for CIPN
* Physical Therapy Examination indicates use of Rebuilder for CIPN
* At least 18 years of age
* Signed informed consent for study population
* Willingness to complete study according to protocol

Exclusion Criteria:

* Patients who do not have CIPN
* Patients <18 years of age
* Inability to or unwilling to sign informed consent
* Unable to read and understand the English language
* Preexisting sensory peripheral neuropathy from other comorbid conditions such as diabetes or alcoholism
* More than three (3) prior ReBuilder treatments; OR ReBuilder within the last 30 days, for sensory peripheral neuropathy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer and chemotherapy induced peripheral neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Changes in touch and sensory by way of change in the Semmes-Weinstein Monofilament Testing | one year
Changes in touch and sensory by way of changes in Functional Gait Assessment | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Regional Medical Center, Philadelphia, Pennsylvania, United States